CLINICAL TRIAL: NCT06741059
Title: Determining the Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Pain and Menstrual Symptoms in Primary Dysmenorrhea
Brief Title: Effect of TENS on Pain and Symptoms in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, ESRA ÜNAL, Dr, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OKU-SBF-EU-01
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Dysmenorrhea
Keywords: Primary Dysmenorrhea; Transcutaneous Electric Nerve Stimulation; Menstrual Pain; nursing
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: This design allows for direct comparison of the active intervention, placebo, and no intervention (control), evaluating the impact of the treatment on the outcomes.
Who Masked: Participant
Masking Description: Study Design: This study follows a parallel design with three groups:
  Experimental Group: Participants in this group receive the active intervention (e.g., Transcutaneous Electrical Nerve Stimulation - TENS).
  Placebo Group: Participants in this group receive a placebo treatment (e.g., a sham TENS treatment or a non-active intervention).
  Control Group: Participants in this group receive no intervention or the standard treatment.
  Blinding: A single-blind design is used in this study, meaning only the participants do not know which group they are assigned to. The research team is aware of the group assignments. This approach helps prevent the participants' expectations from influencing the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The group receiving the TENS treatment (Experimental): The group has received the TENS treatment.
  Interventions: Other: Transkutanöz Elektriksel Sinir Stimülasyonu - TENS
- Placebo Comparator (Placebo Comparator): It is the placebo group where the TENS device is applied, but no treatment is given.
  Interventions: Other: Transkutanöz Elektriksel Sinir Stimülasyonu - TENS
- Control Group (No Intervention): It is the control group, which receives no intervention or standard treatment.

INTERVENTIONS:
Other: Transkutanöz Elektriksel Sinir Stimülasyonu - TENS — Transcutaneous Electrical Nerve Stimulation (TENS) has gained popularity in recent years as a non-invasive method for pain management. TENS works by modulating nerve stimulation through low-frequency electrical currents applied to the skin, reducing pain perception. Its potential effectiveness in alleviating menstrual pain has drawn increasing attention as an alternative treatment option
  Arms: Placebo Comparator; The group receiving the TENS treatment

SUMMARY:
The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Pain and Menstrual Symptoms in Primary Dysmenorrhea

This study aims to investigate the effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) in managing pain and alleviating menstrual symptoms in individuals with primary dysmenorrhea. Primary dysmenorrhea is characterized by severe menstrual pain and accompanying symptoms that negatively impact the quality of life and daily functioning. TENS, a non-invasive and drug-free method, is applied to relieve pain by stimulating nerves through electrical impulses. This research evaluates the impact of TENS on both the intensity of menstrual pain and associated symptoms, offering insights into its potential as an alternative or complementary therapeutic approach.

DETAILED DESCRIPTION:
The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Pain and Menstrual Symptoms in Primary Dysmenorrhea

Primary dysmenorrhea is a common health problem experienced by women during their menstrual periods, significantly affecting their quality of life. It is often characterized by severe abdominal pain, cramp-like symptoms, nausea, headaches, and fatigue. These symptoms can impact social and functional activities, and in some cases, restrict participation in daily routines.

The treatment of primary dysmenorrhea aims to alleviate symptoms and help women experience a more comfortable menstrual period. Traditional treatments include pain relievers, hormonal therapies, and lifestyle changes. However, these methods may not always be sufficient, or some women may avoid them due to potential side effects.

Transcutaneous Electrical Nerve Stimulation (TENS) has gained popularity in recent years as a non-invasive method for pain management. TENS works by modulating nerve stimulation through low-frequency electrical currents applied to the skin, reducing pain perception. Its potential effectiveness in alleviating menstrual pain has drawn increasing attention as an alternative treatment option.

This study aims to evaluate the effects of TENS on pain and menstrual symptoms in women with primary dysmenorrhea. The research will assess the potential of TENS to reduce menstrual pain and compare its effectiveness with other treatment options. If TENS proves to be effective in managing dysmenorrhea symptoms, it could enhance women's quality of life and provide a valuable non-pharmacological treatment alternative.

The findings of this study could contribute to understanding the role of TENS in alleviating dysmenorrhea symptoms and developing effective treatment strategies to improve women's quality of life during their menstrual periods.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Have regular menstrual cycles (lasting 3 to 8 days, with a menstrual cycle range of 21 to 35 days)
* Have dysmenorrhea pain severity rated 4 or higher on the Visual Analog Scale (VAS)

Exclusion Criteria: Women with the following conditions were excluded from the study:

* Secondary dysmenorrhea
* Using oral contraceptives
* Having impaired tissue integrity in the abdominal area
* Having previous experience with TENS
* Having a history of nerve damage or sensory loss
* Having a pacemaker
* Having any systemic diseases
* Being pregnant or in the postpartum period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 93 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous Electrical Nerve Stimulation | 3 months
  Transcutaneous Electrical Nerve Stimulation (TENS) is effective in pain management in women with primary dysmenorrhea. The Visual Analog Scale is a scale where the patient can mark their own pain on a ruler that can be used horizontally or vertically, where the pain is evaluated between 0-10. VCS is used to evaluate both the severity of pain and the effectiveness of the treatment/intervention on pain in various populations. An increase in the score indicates an increase in pain.

SECONDARY OUTCOMES:
Transcutaneous Electrical Nerve Stimulation (TENS) is effective in managing menstrual symptoms in women with primary dysmenorrhea. | 3 months
  Transcutaneous Electrical Nerve Stimulation (TENS) is effective in managing menstrual symptoms in women with primary dysmenorrhea.A scale was developed by Taylor in 1979 to assess the symptoms and intensity of symptoms that occur during menstruation. The Turkish validity and reliability of the scale was performed by Oskay et al. in 2008. The scale, which contains seventeen items, has no sub-dimensions with each symptom being scored between 0 and 5. An increase in score indicates an increase in the intensity of the symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Ünal, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will share the study results, but individual forms will not be shared because they require patient consent.